CLINICAL TRIAL: NCT02237625
Title: Natural History Study of Adult and Pediatric Patients With Hypophosphatasia
Brief Title: Natural History Study of Patients With Hypophosphatasia (HPP)
Acronym: NatHisHPP
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00049204; Pro00049204 (Other: DUHS IRB)
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Hypophosphatasia
Keywords: Hypophosphatasia; HPP
MeSH Terms: conditions — Hypophosphatasia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 100 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Medical History of HPP Patients: Patient clinical data will be collected related to the diagnosis, onset, progression, treatment course and outcome for patients with HPP.

SUMMARY:
Hypophosphatasia (HPP) is a rare inherited metabolic disorder characterized by defective bone and teeth mineralization caused by mutations of the ALPL gene, which encodes for the tissue-nonspecific alkaline phosphatase (TNSALP) isozyme, resulting in decreased serum and bone alkaline phosphatase levels. To date, over 250 different mutations in the gene encoding TNSALP have been associated with HPP. Clinically, the loss of TNSALP function results in progressive skeletal impact as well as progressive impact on all other major organ systems. It clinically manifests as rickets in infants and children and osteomalacia at all ages. The severe form of the disease has been estimated to have a prevalence of about 1 in every 100,000 live births.

DETAILED DESCRIPTION:
Inheritance can be autosomal recessive or dominant, and penetrance is variable resulting in a wide range of clinical expressivity, with a spectrum ranging from stillbirth without mineralized bone to early loss of teeth without bone symptoms. Depending on the age at diagnosis six clinical forms are currently recognized: perinatal (lethal), perinatal benign, infantile, childhood, adult and odontohypophosphatasia. Severe forms of HPP (perinatal and infantile) are inherited as an autosomal recessive trait and in milder forms (adult and odontohypophosphatasia) autosomal recessive and autosomal dominant inheritance coexist.

Because of the rarity of HPP as well as the side spectrum of both clinical presentation and inheritance patterns of the HPP trait, a natural history study cataloging specific clinical data with HPP would prove invaluable for future research into this disease. Specifically, it is our goal to create a comprehensive multi-discipline modality for care for hypophosphatasia patients, researching clinical manifestations of the disease such as extent of bone disease, ophthalmologic manifestations, orthopedic issues, renal issues, musculoskeletal manifestations as well as other more anecdotal findings such as those seen with cochlear implant failures and/or early menopause.

ELIGIBILITY:
Inclusion Criteria:

* Patients or their legal representative must provide written informed consent or, if applicable, qualify for waiver of consent.
* Patients must have a pre-established clinical diagnosis of HPP, as indicated by one or more of the following:

  * Serum alkaline phosphatase (ALP) below the age-adjusted normal range
  * Plasma PLP at least twice the upper limit of normal (no vitamin B6 administered for at least 1 week prior to determination)
  * Evidence of osteopenia or osteomalacia on skeletal radiographs
  * Genetic analysis fof the ALPL gene
* Must be current patient in the Duke University System.

Exclusion Criteria:

* Any patient without confirmation of clinical diagnosis of HPP.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 100 minor and 100 adult subjects will be enrolled into this natural history study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-09; Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Medical History of HPP Patients | 100 years
  Patient clinical data will be collected related to the diagnosis, onset, progression, treatment course and outcome for patients with HPP

SECONDARY OUTCOMES:
long-term efficacy of treatment modalities | 100 years
potential long term complications of the disease and/or treatment | 100 years
quality of life issues for patients living with hypophosphatasia | 100 years

CONTACTS AND LOCATIONS:
Overall Officials: Priya Kishnani, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States